CLINICAL TRIAL: NCT02004366
Title: Linagliptin Inpatient Trial: A Randomized Controlled Trial on the Safety and Efficacy of Linagliptin (Tradjenta®) Therapy for the Inpatient Management of General Surgery Patients With Type 2 Diabetes
Brief Title: Linagliptin Inpatient Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Boston Medical Center (Other); Rush University (Other); University of Denver (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00066548
Record Dates: First submitted 2013-11-19; First posted 2013-12-09 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Linagliptin; hospital hyperglycemia; inpatient diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Linagliptin; Insulin Glargine; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Linagliptin In-hospital (Experimental): Linagliptin once daily+ correction doses of aspart or lispro if needed
  Interventions: Drug: Linagliptin
- Basal Bolus In-hospital (Active Comparator): Glargine once daily and rapid-acting insulin before meals + correction doses of aspart or lispro if needed
  Interventions: Drug: Basal Bolus
- Linagliptin on discharge (Experimental): Patients with admission A1C < 7% will be discharged on same pharmacologic regimen (oral agents, insulin therapy) or linagliptin 5 mg/day. If contraindication to oral anti-diabetics (OAD), discharge patient on linagliptin once daily.
  Interventions: Drug: Linagliptin
- Linagliptin+50%Glargine dose on d/c (Experimental): Patients with admission HbA1c between 7% and 9% will be discharged on previous oral anti-diabetic agents plus linagliptin, and consider glargine insulin at 50% of daily hospital dose. Patient who did not receive glargine in the hospital, discharge on previous OAD + linagliptin once daily, and consider starting glargine at 0.15 unit/kg/day.
  Interventions: Drug: Linagliptin + 50% Glargine dose on discharge
- Linagliptin+80%Glargine dose on d/c (Experimental): Patients with admission HbA1c ≥ 9% will be discharged on previous oral anti-diabetic agents plus linagliptin, and consider glargine insulin at 80% of daily hospital dose. Patient who did not receive glargine in the hospital, discharge on previous OAD + linagliptin once daily, and consider starting glargine at 0.15 unit/kg/day.
  Interventions: Drug: Linagliptin + 80% Glargine

INTERVENTIONS:
Drug: Linagliptin — Linagliptin once daily + correction doses of rapid acting insulin if needed
  Other Names: Tradjenta
  Arms: Linagliptin In-hospital
Drug: Basal Bolus — Basal bolus regimen with glargine once daily and rapid-acting insulin (lispro or aspart) before meals + + correction doses of rapid acting insulin if needed
  Other Names: Glargine (Lantus) + aspart (Novolog) or lispro (Humalog)
  Arms: Basal Bolus In-hospital
Drug: Linagliptin — Patients with admission A1C < 7% will be discharged on same pharmacologic regimen (oral agents, insulin therapy) or linagliptin 5 mg/day for 3 months.
  Other Names: Trajenta
  Arms: Linagliptin on discharge
Drug: Linagliptin + 50% Glargine dose on discharge — Patients with admission HbA1c between 7% and 9% will be discharged on previous oral anti-diabetic agents plus linagliptin, and consider glargine insulin at 50% of daily hospital dose for 3 months.
  Other Names: Trajenta, Lantus
  Arms: Linagliptin+50%Glargine dose on d/c
Drug: Linagliptin + 80% Glargine — Patients with admission HbA1c ≥ 9% will be discharged on previous oral anti-diabetic agents plus linagliptin, and consider glargine insulin at 80% of daily hospital dose for 3 months.
  Other Names: Trajenta, Lantus
  Arms: Linagliptin+80%Glargine dose on d/c

SUMMARY:
This study is a prospective, randomized, open label trial to compare the safety and efficacy of linagliptin (an oral anti diabetic medication) given orally once daily to an insulin regimen of glargine once daily plus rapid-acting insulin before meals. Both of these treatment groups will be given corrective doses of rapid-acting insulin analogs (aspart, lispro or glulisine) before meals if their blood sugars are > 140 mg/dl.

The patients will be monitored for their blood sugars while the hospital.

If patients are agreeable to participate in the discharge part of the study, the investigators will randomized them to a treatment group based on their admission HbA1c. The investigators will follow these patients for 3 months with phone calls and clinic visits, and will monitor their blood sugars. This is to compare the efficacy of linagliptin and our discharge treatment algorithm in controlling blood sugars as out patients.

DETAILED DESCRIPTION:
Specific Aim 1: To determine whether in-hospital glycemic control, as measured by mean daily glucose concentration and frequency of hypoglycemic events, is different between treatment with linagliptin (Tradjenta®) plus correction doses with a rapid-acting insulin analog before meals and a basal bolus regimen with glargine once daily and rapid-acting insulin analog before meals in general surgery patients with T2D.

Specific Aim 2: To determine the efficacy and safety of an A1C based discharge algorithm in controlling BG after discharge in patients with T2D. Patients who participate in the in-hospital arm (Aim 1) will be invited to enroll in this open label prospective outpatient study. The total duration of the study is 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Males or female surgical non-ICU patients ages between18 and 80 years
2. A known history of T2D > 1 month, receiving either diet alone, oral antidiabetic agents: sulfonylureas and metformin as monotherapy or in combination therapy (excluding DPP-4 inhibitors) or low-dose (≤ 0.5 units/kg/day) insulin therapy.
3. Subjects with a BG >140 mg and < 400 mg/dL at time of randomization without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 mEq/L or positive serum or urinary ketones)

Exclusion Criteria:

1. Age < 18 or > 80 years.
2. Subjects with increased BG concentration, but without a history of diabetes (stress hyperglycemia).
3. Subjects with a history of type 1 diabetes (suggested by BMI < 25 requiring insulin therapy or with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria) (43).
4. Treatment with dipeptidyl peptidase-4 (DPP4) inhibitor or Glucagon-like peptide-1 (GLP1) analogs during the past 3 months prior to admission.
5. Acute critical illness or coronary artery bypass graft (CABG) surgery expected to require admission to a critical care unit.
6. Subjects with gastrointestinal obstruction or adynamic ileus or those expected to require gastrointestinal suction.
7. Patients with clinically relevant pancreatic or gallbladder disease.
8. Patients with previous history of pancreatitis
9. Patients with acute myocardial infarction, clinically significant hepatic disease or significantly impaired renal function (GFR < 30 ml/min).
10. Chronic use of steroid with total daily dose (prednisone equivalent) >5 mg/day
11. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
12. Pregnancy or breast feeding at time of enrollment into the study.
13. Patients who received supplemental sliding scale insulin >72 hours prior to randomization
14. Patients who received basal insulin > 48 hours prior to randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, Principal Investigator — Emory University SOM
Locations (5):
- United States (5):
  - University of Colorado, Denver, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between February 2014 and October 2016. Patients who participated in the in-hospital study period were invited to enroll in the prospective outpatient study. Of 250 in-patient participants, 224 accepted enrollment into outpatient study.
Pre-assignment Details: Of the 295 subjects consented, there were 15 screen failures. 30 (out of remaining 280 patients) were excluded from participation: 11 patients stayed <24 hours, 1 patient received corticosteroids, and 18 patients didn't receive medication. Therefore, 250 patients started the study.
Groups:
- Linagliptin In-hospital: Linagliptin once daily + correction doses of aspart or lispro if needed.
  Linagliptin: Linagliptin once daily + correction doses of rapid acting insulin if needed
Period: In-hospital
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Started | 128 | 122 | 0 | 0 | 0
Completed | 128 | 122 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: On Discharge
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Started | 0 | 0 | 92 | 93 | 39
Completed | 0 | 0 | 92 | 93 | 39
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants are represented for the two stages of the study (in-hospital and discharge), and are counted more than once in the Total.
Groups:
- Total: Total of all reporting groups
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c | Total
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39 | 474
Age, Continuous [Mean (Standard Deviation); unit: years]
  In-hospital | 58 (11) | 58 (12) | NA (NA) — Arms are not relevant to the named period | NA (NA) — Arms are not relevant to the named period | NA (NA) — Arms are not relevant to the named period | 57.8 (11.3)
  Discharge | NA (NA) — Arms are not relevant to the named period | NA (NA) — Arms are not relevant to the named period | 58.8 (10.0) | 57.1 (11.7) | 50.7 (11.5) | 56.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  In-hospital: Female | 66 | 58 | NA — Arms are not relevant to the named period | NA — Arms are not relevant to the named period | NA — Arms are not relevant to the named period | NA — Total not calculated because data are not available (NA) in one or more arms.
  In-hospital: Male | 62 | 64 | NA — Arms are not relevant to the named period | NA — Arms are not relevant to the named period | NA — Arms are not relevant to the named period | NA — Total not calculated because data are not available (NA) in one or more arms.
  Discharge: Female | NA — Arms are not relevant to the named period | NA — Arms are not relevant to the named period | 54 | 49 | 7 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Discharge: Male | NA — Arms are not relevant to the named period | NA — Arms are not relevant to the named period | 38 | 44 | 32 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  In-hospital Black | 59 | 58 | 0 | 0 | 0 | 117
  In-hospital White | 44 | 46 | 0 | 0 | 0 | 90
  In-hospital Hispanic | 21 | 12 | 0 | 0 | 0 | 33
  In-hospital Other | 4 | 6 | 0 | 0 | 0 | 10
  Discharge Black | 0 | 0 | 42 | 46 | 23 | 111
  Discharge White | 0 | 0 | 36 | 33 | 6 | 75
  Discharge Hispanic | 0 | 0 | 13 | 10 | 5 | 28
  Discharge Other | 0 | 0 | 1 | 2 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States: In-hospital | 128 | 122 | 0 | 0 | 0 | 250
  United States: Discharged | 0 | 0 | 92 | 93 | 39 | 224

OUTCOME MEASURES:

1. Primary Outcome: Differences in Glycemic Control
Description: Determine differences in glycemic control as measured by mean daily BG concentration between linagliptin alone and basal bolus therapy group.
Time Frame: Inpatient (average 5 days) and outpatient up to 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
mg/dl | 171 (47) | 159 (41) | 126 (22) | 132 (28) | 142 (24)

2. Secondary Outcome: Hypoglycemia <70 mg/dl
Description: Subjects with Hypoglycemia <70 mg/dl
Time Frame: Inpatient (average 5 days) and outpatient up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
Participants | 2 | 14 | 8 | 15 | 10

3. Secondary Outcome: Hyperglycemia
Description: Subjects with BG > 300 mg/dl
Time Frame: Inpatient (average 5 days) and outpatient up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
Participants | 22 | 18 | 6 | 11 | 7

4. Secondary Outcome: Daily Dose of Insulin
Description: Total daily dose of insulin
Time Frame: Inpatient (average 5 days) and outpatient up to 12 weeks
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
units/kg/day | 0.09 (0.17) | 0.31 (0.15) | 0.23 (0.1) | 0.18 (0.1) | 0.24 (0.1)

5. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay (ONLY for inpatient arms 1 and 2)
Time Frame: During Hospitalization
Population: Length of hospital stay is applicable ONLY for inpatient arms (1 and 2)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 0 | 0 | 0
Days | 4 [3 to 5] | 3 [3 to 6] |  |  |

6. Secondary Outcome: Number of Participants Requiring ICU Care During Hospitalization
Description: Need for intensive care unit (ICU) care (transfer to ICU) during hospitalization
Time Frame: During Hospitalization-average 5 days
Population: Transfer to ICU is applicable ONLY for inpatient arms (1 and 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 0 | 0 | 0
Participants | 1 | 0 | 0 | 0 | 0

7. Secondary Outcome: Hospital Complications
Description: Subjects with composite complication (ONLY for inpatient arms 1 and 2)
Time Frame: During Hospitalization-average 5 days
Population: Composite complication during hospitalization is applicable ONLY for inpatient arms (1 and 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 0 | 0 | 0
Participants | 14 | 11 |  |  |

8. Secondary Outcome: Acute Renal Failure During Hospitalization
Description: Subjects with Acute renal failure (ONLY for inpatient arms 1 and 2)
Time Frame: During Hospitalization-average 5 days
Population: Acute renal failure during hospitalization is applicable ONLY for inpatient arms (1 and 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 0 | 0 | 0
Participants | 6 | 4 |  |  |

9. Secondary Outcome: Hospital Mortality
Description: Hospital mortality (ONLY in-patient). Mortality is defined as death occurring during hospital stay.
Time Frame: During Hospitalization-average 5 days
Population: Hospital mortality is applicable ONLY for inpatients arms (1 and 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 0 | 0 | 0
Participants | 0 | 0 |  |  |

10. Secondary Outcome: Fasting BG Concentration
Description: Average - per hospital stay - fasting BG concentration (for in-hospital groups), and average - per outpatient follow-up period - fasting BG concentration (for discharge groups)
Time Frame: During Hospitalization (average 5 days) and outpatient up to 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
mg/dl | 160 (44) | 167 (44) | 125 (22) | 133 (27) | 141 (25)

11. Secondary Outcome: Subjects With Wound and Other Infections
Description: Subjects with wound and other infections.
Time Frame: During Hospitalization and outpatient up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
Participants | 7 | 3 | 3 | 5 | 4

12. Secondary Outcome: HbA1c Level
Description: HbA1c level at admission (for in-patient arms) and HbA1c level at 12-week follow-up outpatient visit (for discharge arms).
Time Frame: Admission to the hospital and 12-week follow-up outpatient visit
Measure: Mean (Standard Deviation); unit: % DCCT
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
% DCCT | 7.6 (1.9) | 8.0 (2.0) | 6.6 (0.8) | 7.0 (1.0) | 8.6 (2.7)

13. Secondary Outcome: Hypoglycemia < 40 mg/dl
Description: Subjects with Hypoglycemia < 40 mg/dl
Time Frame: Inpatient and up to 12 weeks outpatient
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
Participants | 1 | 0 | 1 | 0 | 1

14. Secondary Outcome: Emergency Room Visits
Description: Number of ER visits ONLY for outpatient arms 3,4, and 5.
Time Frame: 3 months after discharge
Population: Emergency visits reported only for outpatient time. Inpatient (hospital) patients cannot have ER visits
Measure: Number; unit: Visits
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 0 | 0 | 92 | 93 | 39
Visits |  |  | 11 | 11 | 9

15. Secondary Outcome: Subjects With Surgical Reinterventions
Description: Subjects with surgical re-interventions.
Time Frame: Inpatient and up to 12 weeks outpatient
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 128 | 122 | 92 | 93 | 39
Participants | 6 | 4 | 5 | 3 | 3

16. Secondary Outcome: Outpatient Mortality
Description: Deaths among patients after hospital discharge.
Time Frame: 3 months after discharge
Population: Deaths after hospital discharge are applicable ONLY for outpatient arms (3, 4 and 5).
Measure: Count of Participants; unit: Participants
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
Number analyzed (Participants) | 0 | 0 | 92 | 93 | 39
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 weeks (average 5 days in hospital and 12 weeks after discharge)
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Arm/Group | Linagliptin In-hospital | Basal Bolus In-hospital | Linagliptin on Discharge | Linagliptin+50%Glargine Dose on d/c | Linagliptin+80%Glargine Dose on d/c
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/122 | 0/92 | 0/93 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/128 | 0/122 | 12/92 | 14/93 | 9/39
Other Adverse Events (participants affected / at risk) | 25/128 | 15/122 | 3/92 | 1/93 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linagliptin In-hospital (N=128) | Basal Bolus In-hospital (N=122) | Linagliptin on Discharge (N=92) | Linagliptin+50%Glargine Dose on d/c (N=93) | Linagliptin+80%Glargine Dose on d/c (N=39)
ICU admission (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Resurgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 5 (5) | 3 (7) | 3 (3)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 5 (6) | 4 (4)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Genitourinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linagliptin In-hospital (N=128) | Basal Bolus In-hospital (N=122) | Linagliptin on Discharge (N=92) | Linagliptin+50%Glargine Dose on d/c (N=93) | Linagliptin+80%Glargine Dose on d/c (N=39)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hematologic (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical Reintervention (Surgical and medical procedures) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Renal (Renal and urinary disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Infections (Infections and infestations) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT02004366/Prot_SAP_000.pdf